CLINICAL TRIAL: NCT04250532
Title: Pulse Oximetry in Healthy SubjEcts ImmergeD in OceaN.
Acronym: POSEIDON
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/48
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Drowning
MeSH Terms: conditions — Drowning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lifeguard: Lifeguards who work on the Atlantic coast of Gironde France.
  Interventions: Other: Drowning

INTERVENTIONS:
Other: Drowning — Measurement of pulse oximetry, after lifeguard immersion during their morning training

SUMMARY:
Drowning is the 3rd leading cause of accidental death in the world. One of the tools used by lifeguards to help ER assess gravity, is pulse oximetry. Its measure is variable even in optimal condition and its accuracy can be altered by factors specific to the patient and by environmental factors. The conditions gathered during a drowning rescue are thus propitious to a misleading evaluation. Assessing its reliability and looking for influencing factors of the measure of pulse oximetry could help for pre-hospital care management.

DETAILED DESCRIPTION:
The research focuses on the measurement of pulse oximetry among lifeguard on the Atlantic coast of Gironde, France, before and after their daily training, using a standardized measurement protocol.

The follow-up will be done during the beach monitoring period during the summer of 2020. A total of 3 months of measurement collection is expected.

ELIGIBILITY:
Inclusion Criteria:

* Lifeguard working on the Girondine Atlantic coast
* up to 18 years old,
* no smoker,
* No chronic pathology.

Exclusion Criteria:

* Chronic cardiac pathology,
* Chronic respiratory pathology,
* Acrosyndrome,
* Smoker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lifeguards working on the Girondine Atlantic coast
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of abnormal pulse oximetry measure | 3 months after inclusion day
  Quantify the number of subjects, whose pulse oximetry is measured as abnormal (superior to 94%) after immersion for 15 min in the ocean, in real condition.

SECONDARY OUTCOMES:
Variation of pulse oximetry according to individuals factors | 3 months after inclusion day
  Measures of immersion time, BMI before / after immersion.
Variation of pulse oximetry according to environnementals factors | 3 months after inclusion day
  Measures of air, water temperatures, felt air temperature, wet thermometer temperature, wind speed before / after immersion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No